CLINICAL TRIAL: NCT01190137
Title: Bio-equivalency Study of the Effects of Vitamin D2 and Vitamin D3 Supplements on 25-hydroxyvitamin D Levels in Exclusively Breast Fed Canadian Infants
Brief Title: Study Comparing Two Isoforms of Vitamin D Supplements for Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Principal Investigator, Hope Weiler, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A09-M108-09A
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Optimal vitamin D status; 25-hydroxy vitamin D; Rickets and bone mineralization; Breast fed infants; Cholecalciferol and ergocalciferol
MeSH Terms: conditions — Rickets; Breast Feeding | interventions — Cholecalciferol; Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 400 IU Vitamin D3 (Active Comparator)
  Interventions: Dietary Supplement: Cholecalciferol (D3) or ergocalciferol (D2)
- 400 IU Vitamin D2 (Experimental)
  Interventions: Dietary Supplement: Cholecalciferol (D3) or ergocalciferol (D2)

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (D3) or ergocalciferol (D2) — 400 IU administered as 1 drop daily for 3 months
  Other Names: Baby D Drops

SUMMARY:
There are two different types of vitamin D - vitamin D3 (animal source) and vitamin D2 (plant source). Almost all the usual vitamin D preparations for infants available in Canadian pharmacies contain vitamin D3 which may not be suitable for families who avoid animal products for social or religious reasons. The purpose of this study is to learn more about the two forms of vitamin D and if blood levels of vitamin D are similar in infants after taking them. Forty-eight breastfed infants will be randomly assigned to 400 IU of either vitamin D2 or D3 supplement for 3 months starting at 1 month of age. The difference in blood vitamin D levels, after 3 months of supplementation, between the two groups will help determine if the two supplements are equal.

DETAILED DESCRIPTION:
Vitamin D is important to develop strong bones and teeth as well as to prevent rickets, a childhood bone disease in which the bones get very soft and bend. the investigators know that vitamin D can be produced by cells in our skin during sunny months of the year but there is a concern about the safety of sun exposure in infants. As well breast milk contains very little vitamin D. It is for this reason that Health Canada recommends all breast fed babies should receive 400 IU of vitamin D per day. There are two different types of vitamin D - vitamin D3 (animal source) and vitamin D2 (plant source). Standard infant preparations in Canada tend to be in the vitamin D3 form. To date, there is insufficient information to judge the equivalency of 400 IU of vitamin D2 and D3 given daily in very young Canadian infants. In view of over 1 million Canadian families practicing vegetarianism, this would appear to be an important and not yet answered question. The investigators cannot extrapolate from the adult data because the infant physiology is immature relative to adults and absorption, especially of fat soluble vitamins differs. This area needs to be better evaluated to emphasize the optimal isoform of vitamin D during infancy necessary for the development of adequate bone mass.

This study aims to compare the relative ability of equal daily intakes of vitamin D2 and D3, amounts (400 IU/d) currently recommended by Health Canada, to support circulating 25(OH)D concentrations after 3 months of supplementation in breastfed newborns. In particular, whether both supplements are equally effective in their ability to achieve and sustain optimal plasma 25(OH)D concentrations, defined as 25(OH)D values between 75-225 nmol/L.

Design: Randomized clinical trial in which 48, 1 month old infants, will be randomized to either the vitamin D2 or D3 isoform at the standard of care dosage (400 IU daily) for 3 months; a sufficient time to observe a change of vitamin D status ascribed to the supplement. Infant physiology is immature and evolving and the time to stabilize 25-hydroxy vitamin D (25(OH)D) is approximately 3 weeks (half-life). Supplements will be double blinded to participants, investigators and all staff.

Recruitment: Infants will be recruited from 1 large primary care center located in the greater Montreal area. The goal is for infants to begin the study at 4 weeks of age but a range of +/- 2 weeks. Rolling recruitment over a 9 months period with a 3 month follow-up for all beginning in May 2010. This covers both the synthesizing and non synthesizing periods of vitamin D. This age group has been selected (first month of life) since vitamin D stores transferred from the mother begin to decrease owing to the 15 to 30 day half life of 25(OH)D. After this point, infants need a source of vitamin D other than breast milk or sunshine. Because the majority of Canadian infants are now breastfed for at least 3-6 months of age the first 4 months of life appear to be an important time frame to examine the relative potency of the 2 isoforms.

Frequency and duration of follow up: Infants will be followed for 3 months with 2 visits, at baseline (~1 month) and the end of the study (~4 months). Visits will include anthropometric assessment and blood collection for the assessment of 25(OH)D and parathyroid hormone (PTH) concentrations. Bottles of supplement will be weighed upon receipt and return for compliance. As well, parents will be asked to self-report compliance at each visit. In order to encourage continued supplementation during the 3 month intervention, the investigators plan to a schedule a reminder phone call at approximately 1½ months post the baseline visit. Vitamin D supplementation of infants prior to the initial visit (birth to visit 1) will be documented, but considered as systematic error. Maternal baseline information will be collected at the first visit including demographics, ethnicity, pregnancy history and sun exposure during pregnancy. This data will be used to characterize the study population. At each visit, the health status and sun exposure and sunscreen use of the infants will be assessed. A computerized narrow band reflectometer will be utilized to measure skin pigmentation on unexposed skin of the inner upper arm and forehead. Procedures will be performed using guidelines established by the European Society of Contact Dermatitis. This test estimates melanin content of the skin which influences vitamin D status.

Sample procurement: At both visits, blood will be collected from infants using a capillary blood sample and from mothers by venipuncture. All samples will be taken between 8 and 10 am to control for diurnal variation. Approximately 1 ml of heparinized blood will be collected from infants via heel/finger prick and 5 ml from mothers.

Plasma 25(OH)D and PTH concentrations: Response to supplementation will be evaluated by the change in plasma 25(OH)D and PTH. Mothers 25(OH)D status will also be obtained to determine that both groups are similar as mother's vitamin D status can affect infant's vitamin stores and risk of hypovitaminosis. Mother's vitamin D status will also allow us to better establish total infant vitamin D exposure through maternal placental transfer of vitamin D. If there is no change, the proportion with 25(OH)D below target will be examined. Both vitamin D and PTH will be measured using an automated chemiluminescent assay system (Liaison, Diasorin). All analyses will be completed in a laboratory meeting the performance targets set by the Vitamin D External Quality Assessment Scheme (DEQAS).

Anthropometry: Infant's weight, length and head circumference will be taken at each visit. Gestational age will be documented from the vaccination booklet. Growth will be assessed using triplicate measurements of weight (to nearest g without clothing/diaper using a digital infant scale) and head circumference (to the nearest 0.1 cm using non-stretchable tape). Data will be expressed in absolute units and z-scores using data from the World Health Organization growth charts at each age. Mother's weight, height and body composition (% body fat using bioelectrical impendence will be measured to accurately describe the population.

Infant nutrition: Information of infant feeding status (exclusively, predominately breastfed or formula fed) will be collected at each visit as well as the reminder telephone call (approximately 1½ most post supplementation). If formula is consumed, information about specific amounts consumed, frequency, brands as well as additional multivitamins/minerals will also be collected.

Mother's nutrition: Mother's vitamin D intake from diet and supplements will be assessed during lactation using a 24 hour recall, using the US Department of Agriculture 5-step multiple-pass method for dietary recall, conducted with a registered dietitian at each visit. The correct assessment of 25(OH)D from dietary food records is limited as current food sources of vitamin D (such as fish) are consumed weekly or a few times/month. 24-hours recalls will likely miss important food sources thus, the Canadian adapted Harvard Food Frequency Questionnaire will be completed to assess last 3 months of usual food intake.

Safety: Participants found to be below the optimal range of vitamin D [25(OH)D ≤ 75 nmol/L, 30 ng/ml] or any value exceeding 225 nmol/L [90 ng/ml] after the 3-month supplementation period, upon participant consent, will be contacted and referred to their pediatrician for appropriate treatment. If permitted by the participant, the physician will be contacted directly with the results. Both maternal and infant 25(OH)D values collected at the visit 2 will be made available to all participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, singleton term infants of appropriate for gestational age, according to Centers for Disease Control (CDC) growth charts based on weight at birth between 5th and 95th percentiles for sex
* Born to healthy breastfeeding women
* Exclusively breast fed infants from birth, according to WHO definition: breast milk, expressed breast milk, vitamins, minerals and medicine but not including water, breast milk substitutes, other liquids and solid foods.

Exclusion Criteria:

* Infants of mothers with a history of gestational diabetes or hypertension in pregnancy; chronic alcohol use; malabsorption syndromes (Celiac disease, Crohn's, etc.), due to malabsorption of fat soluble vitamins
* Mothers taking any medications that can affect vitamin D metabolism (anticonvulsants and corticosteroids)
* Mothers taking ≥ 2,000 IU/d of vitamin D from supplementation

Ages: 2 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Equivalency of isoforms | 3 months
  To compare the relative ability of daily oral supplementation of 400 IU in the form of vitamin D3 or D2 to achieve and sustain optimal plasma 25(OH)D concentrations, defined as 25(OH)D values between 75-225 nmol/L, in exclusively breastfed infants.

CONTACTS AND LOCATIONS:
Overall Officials: Hope A, Weiler, PhD, RD, Principal Investigator — McGill University; Celia Rodd, MD, Principal Investigator — Montreal Children's Hospital, McGill University Health Center; Sina Gallo, MSc, RD, Principal Investigator — McGill University
Locations (1):
- Mary Emily Clinical Nutrition Research Unit, Ste. Anne de Bellevue, Quebec, Canada

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Gallo S, Phan A, Vanstone CA, Rodd C, Weiler HA. The change in plasma 25-hydroxyvitamin D did not differ between breast-fed infants that received a daily supplement of ergocalciferol or cholecalciferol for 3 months. J Nutr. 2013 Feb;143(2):148-53. doi: 10.3945/jn.112.167858. Epub 2012 Dec 19. PMID 23256143